CLINICAL TRIAL: NCT03634917
Title: Investigation of the Efficacy of Acamprosate and Calcium in Comparison to Placebo as Validation of a Behavioural Test for Alcohol Dependence (TEMACA)
Brief Title: Investigation of the Efficacy of Acamprosate and Calcium in Comparison to Placebo as Validation of a Behavioural Test for Alcohol Dependence
Acronym: TEMACA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TUD-TEMACA-069
Record Dates: First submitted 2018-07-25; First posted 2018-08-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Alcoholism
Keywords: Acamprosate; Calcium; alcohol self-administration
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Calcium Carbonate; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acamprosate (Active Comparator): 1 capsule with Acamprosate calcium
  * oral use
  * 3 times / day (morning, noon, evening)
  * 666 mg per capsule
  * 14 - 19 days
  Interventions: Drug: Acamprosate Calcium; Drug: Placebo lead in
- Calcium Carbonate (Active Comparator): 1 capsule with Calcium Carbonate
  * oral use
  * 3 times / day (morning, noon, evening)
  * 1500 mg Calcium Carbonate (= 600 mg Calcium 2+)
  * 14 - 19 days
  Interventions: Drug: Calcium Carbonate; Drug: Placebo lead in
- Placebo (Placebo Comparator): 1 capsule placebo,
  * oral use
  * 3 times / day (morning, noon, evening)
  * 14 - 19 days
  Interventions: Drug: Placebo; Drug: Placebo lead in

INTERVENTIONS:
Drug: Acamprosate Calcium — 1 capsule with 666 mg Acamprosate
  Other Names: Campral
  Arms: Acamprosate
Drug: Calcium Carbonate — 1 capsule with 1500 mg Calcium Carbonate
  Other Names: Calcium
  Arms: Calcium Carbonate
Drug: Placebo — 1 Capsule with Placebo (lactose monohydrate, micro crystalline cellulose, magnesium stearate)
  Arms: Placebo
Drug: Placebo lead in — 1 Capsule with Placebo (lactose monohydrate, micro crystalline cellulose, magnesium stearate)

SUMMARY:
Validation of a Test System to develop new medications for alcoholism (TEMA)

The 'TEMA', a progressive-work alcohol self-administration paradigm, can be validated by reproducing the effect of Acamprosate and prove the effect of Calcium to reduce motivation to work for alcohol after 14 - 19 days of treatment during a period of 15 - 20 days of alcohol abstinence in a randomized, double-blind, placebo-controlled three-arm parallel-group design.

DETAILED DESCRIPTION:
Objective of this study is to show that a laboratory alcohol self-administration method can predict the therapeutic potential of new compounds to reduce relapse in alcohol-dependent patients.

The 'TEMA' translates several animal behavioral paradigms of alcohol self-administration into corresponding human experiments.

84 at least high risky drinkers (WHO) with at least mild alcohol use disorder perform two alcohol self-administration experiments, one before and one after 14-19 days of randomized double-blinded treatment with Acamprosate, Calcium Carbonate or Placebo.

Each alcohol request requires prior work in a constant attention task according to a progressive schedule to earn the next alcohol infusion.

Secondary objectives refer to investigations, whether

1. administration of Acamprosate or Calcium Carbonate in comparison to placebo leads to a change in perception of subjective alcohol effects
2. effectiveness of Acamprosate or Calcium can be predicted by calcium parameters (baseline and changes during medication period)
3. administration of Acamprosate or Calcium leads to a reduction in alcohol craving
4. Frequency of alcohol consumption during the imposed abstinence period differs between treatment groups and influences primary outcome
5. study participation modifies motivation to change drinking habits and utilization of addiction care services
6. Acid sphingomyelinase (ASM) activities are applicable as biomarker and predictor of medication effects.
7. safety issues occur due to study medication

ELIGIBILITY:
Inclusion Criteria:

1. male and female volunteers aged 25 to 55 years, who meet or met the diagnostic criteria of an at least mild alcohol use disorder (DSM-5), but do not want to cease alcohol consumption
2. willingness to stop alcohol and drug consumption for 15-20 days for the purpose of study participation
3. at least high risky alcohol drinkers (WHO) in the Timeline Follow-back Interview over the last 45 day with an average amount of alcohol of 60 g/day (men) or 40 g/day (women) with at least 4 drinking days per week
4. informed consent
5. ability to swallow a placebo capsule
6. not more than 6 consecutive alcohol abstinent days between screening and visit 2

Exclusion Criteria:

1. Current Substance dependence (illegal drugs) ICD-10 or DSM-IV
2. Intention to stop alcohol consumption immediately and permanently
3. Current or previous disease that could cause a clinically relevant hazard (e.g. pancreatitis, cirrhosis)
4. kidney stone disease
5. Current Treatment with psychotropic drugs or current psychiatric disorder in need of treatment
6. alcohol withdrawal symptoms (at Screening, visit 1 or visit 2) with CIWA-Ar-Score > 6 points or arterial blood pressure >160 mm Hg or diastolic blood pressure > 100 mm Hg or heart rate >105 bpm (when breath alcohol concentration 0 mg%)
7. history of epileptic seizure or delirium
8. routine laboratory parameters, indicating relevant liver-, pancreas- or kidney injury, an acute infection, anemia or lack of vitamins (ASAT, ALAT, lipase > threefold of the standard at screening, Quick's value < 70%, creatinine > 120 µmol/l, eGFR < 30 mol/min/1.73 m², leucocytes > 13000/µl, haemoglobin < 7.5 mmol/l (men) or 6.5 mmol/l (women), MCV > 105 fl, calcium level at screening > 2.7 mmol/l
9. body weight > 120 kg (Screening)
10. Breath alcohol concentration at screening or visit 1 or visit 2 two times > 0 mg% or drug screening two times positive for opiate, cannabis, cocaine, amphetamine, benzodiazepine
11. history of hypersensitivity to alcohol or one of the used medicinal products, of their ingredients or medicinal products with similar chemical structures
12. history of inefficient treatment with Acamprosate
13. participation in another clinical trial within the last 4 weeks before inclusion
14. disorders, which will not allow the subject to assess the character and importance or possible consequences of the clinical trial
15. pregnant or breastfeeding women
16. women capable of bearing children, except women who fulfil following criteria:- post-menopausal (12 months natural amenorrhoea or 6 month amenorrhoea and Serum FSH >40 ml U/ml) - post operative (6 weeks after ovariectomy on both sides with or without hysterectomy) - regular and correct use of a contraceptive method with an error Quote of < 1 % per year (for example implants, depot injections, oral contraceptive, IUP). It has to be recognized that a combined oral contraception - in contrast to pure progesterone compounds - have a failure rate of < 1 %. Hormone IUDs with a Pearl Index of 1 % are safer than copper IUDs. - sexual abstinence - vasectomy of the Partner)
17. participant is not expected to comply with the protocol (for example lacking compliance)
18. less than 200 cumulative work trials for alcohol (in constant attention task) on 1st alcohol self-administration day
19. specific contraindications for Acamprosate or Calcium Carbonate (according prescribing information)

    1. hypercalcemia, e.g. due to hyperparathyroidism, overdosage vitamin D, paraneoplastic
    2. renal insufficiency (eGFR < 30ml/min/1.73m²), creatinine >120 µmol/l
20. intake of Vitamin D compounds or cardioactive glycosides

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Difference between cumulative CAT trials for alcohol on 1st alcohol self-administration (ASA) day and 2nd ASA day | 18 to 31 days between 1st and 2nd measurement
  Each alcohol request requires prior work according to a progressive schedule (i.e., runs of the constant attention task) to earn the next alcohol infusion.
  Primary outcome measure is the difference in the cumulative number of work sets for alcohol in the "constant attention task" (CAT) between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5).
  Comparison between:
  1. Acamprosate and Placebo and
  2. Calcium Carbonate and Placebo

SECONDARY OUTCOMES:
Difference between "break points" for alcohol on 1st alcohol self-administration (ASA) day and 2nd ASA day | 18 to 31 day between 1st and 2nd measurement
  The "break point" is the number of the last alcohol request before subjects stop to work for more alcohol.
Difference between max. achieved blood alcohol concentrations (BAC) on 1st alcohol self-administration (ASA) day and 2nd ASA day | 18 to 31 day between 1st and 2nd measurement
  Max. BAC during alcohol self-administration
Difference between cumulative CAT trials for sodium chloride on 1st alcohol self-administration (ASA) day and 2nd ASA day. | 18 to 31 days between 1st and 2nd measurement
  Sodium chloride is an alternative reinforcer on alcohol self-administration.
  Each Sodium chloride request requires prior work according to a progressive schedule (i.e., runs of the constant attention task) to earn the next sodium chloride infusion.
  Outcome measure is the difference in the cumulative number of work sets for sodium chloride (as an alternative reinforce) in the "constant attention task" (CAT) between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5).
Differences in 1st and 2nd half of self-administration periods between cumulative CAT trials for alcohol on 1st alcohol self-administration (ASA) day and 2nd ASA day of 1st and 2nd half of self-administration periods. | 18 to 31 days between 1st and 2nd measurement
  Each alcohol request requires prior work according to a progressive schedule (i.e., runs of the constant attention task) to earn the next alcohol infusion.
  Outcome measure is the difference in the cumulative number of work sets for alcohol in the "constant attention task" (CAT) between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5), considering the 1st and 2nd half of the self-administration period separately
Differences in 1st and 2nd half of self-administration periods between "break points" for alcohol on 1st alcohol self-administration (ASA) day and 2nd ASA day. | 18 to 31 days between 1st and 2nd measurement
  The "break point" is the number of the last alcohol request before subjects stop to work for more alcohol.
  Outcome measure is the the difference in break points for alcohol between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5), considering the 1st and 2nd half of the self-administration period separately.
Differences in 1st and 2nd half of self-administration periods between max. achieved blood alcohol concentrations (BAC) for alcohol on 1st alcohol self-administration (ASA) day and 2nd ASA day. | 18 to 31 days between 1st and 2nd measurement
  Outcome measure is the the difference in max. achieved blood alcohol concentrations between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5), considering the 1st and 2nd half of the self-administration period separately.
Differences in 1st and 2nd half of self-administration periods between cumulative CAT trials for sodium chloride on 1st alcohol self-administration (ASA) day and 2nd ASA day. | 18 to 31 days between 1st and 2nd measurement
  Sodium chloride is an alternative reinforcer on alcohol self-administration.
  Each Sodium chloride request requires prior work according to a progressive schedule (i.e., runs of the constant attention task) to earn the next sodium chloride infusion.
  Outcome measure is the difference in the cumulative number of work sets for sodium chloride in the "constant attention task" (CAT) between first alcohol self-administration day (baseline, without medication, visit 2) and the second alcohol self-administration day (after 14-19 days medication, visit 5), considering the 1st and 2nd half of the self-administration period separately
Differences between subjective alcohol effects on 1st ASA day and 2nd ASA day | 18 to 31 days between 1st and 2nd measurement
  alcohol-induced changes in stimulation, sedation, negative alcohol effects, craving, well-being, subjective feeling of drunkenness, subjective number of drinks and thirst measured with visual analogue scales ("Quizzer") before, 2 x during and after the alcohol infusion period.
  scale ranges: minimum = 0 to maximum = 100
  Higher values on a scale represent an increase of aforementioned subjective alcohol effects.
  Comparison between 1st ASA and 2nd ASA day
Calcium parameters on 1st ASA and 2nd ASA day | 18 to 31 day between 1st and 2nd measurement
  magnesium, phosphate, total calcium, albumin, parathormone, 25-hydroxyvitamin D measurement at baseline and difference between 2nd and 1st ASA
Alcohol craving (OCDS) "Obsessive Compulsive Drinking Scale" (OCDS) | 18 to 31 days between 1st and 2nd measurement
  Craving measured with "Obsessive Compulsive Drinking Scale" (OCDS) before 1st and 2nd ASA The OCDS is a 14-item self-rating instrument. It provides a total and two subscale (1: obsessive, 2. compulsive) scores, that measure aspects of alcohol craving.
Violation of imposed alcohol abstinence | 15-20 days (abstinence period)
  in % of the days with alcohol consumption (measured with timeline follow-back, measured at visit 5)
Readiness to change | 39 - 90 days between screening and visit 6, 6-8 weeks between visit 6 and follow-up
  "Readiness to change" questionnaire 12-item instrument for measuring the "stage of change" at screening, visit 6 and follow-up.
  The test has three four-item subscales to allocate patients to a stage of change: pre-contemplation (P), contemplation (C) or action (A), based on the stages of change model (by Prochaska and DiClementel)
  Answers are given on a scale ranging from 'strongly disagree' ("-2") through "0" to to 'strongly agree' (+2) . The range for each subscale is -8 to +8.
  Each subject is allocated to the stage on which it reached the highest score.
Drinking habits | 39 - 90 days between screening and visit 6, 32 - 55 days between visit 1 and visit 6
  Drinking habits measured with Timeline Follow-back Interview over 45 days before study start (measured at screening) and over the entire study duration (measured at visits 1, 3, 5, 6 and follow-up)
  a) % drinking days, b) average amount of alcohol per drinking day, c) % of binge days (alcohol consumption over 60 g /d (men) or 48 g / d (women)), d) average amount of alcohol per binge day,
utilization of addiction care services | 39 - 90 days between screening and visit 6, 32 - 55 days between visit 1 and visit 6
  does the subject frequent addiction care services at Screening, visit 6 and follow-up
Acid sphingomyelinase (ASM) activities | screening, 18 to 31 day between 1st and 2nd measurement, 2.5 hours from begin to end of ASA
  analysis in serum at screening at visits 2 and 5, before and after alcohol self-administration
Acamprosate blood level | one-time measurement after 14 - 19 days of medication intake (at visit 5)
  measured on 2nd ASA day (visit 5)

OTHER OUTCOMES:
CIWA-Ar-Score | 39 - 90 days between screening and visit 6, 32 - 55 days between visit 1 and visit 6
  Clinical Institute Withdrawal Assessment for Alcohol Scale, revised
  It is a 10-item scale for clinical quantitation of the severity of the alcohol withdrawal syndrome.
  Each item is rated on a scale from 0 to 7, except for "Orientation" which is rated on scale 0 to 4.
  The total CIWA-Ar score is the sum of all 10 items.
  measured at Screening, Visits 1-6.
adverse events / serious adverse events | 32 - 55 days between visit 1 and visit 6
  partially standardized interview about adverse events / serious adverse events
  measured at visits 1-6

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie; Technische Universität Dresden, Dresden, Saxony, Germany

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03634917/SAP_000.pdf